CLINICAL TRIAL: NCT03929341
Title: Risk Evaluation and Stratification of Low Risk for Cardiovascular Disease in Women: An Innovative Strategy for Investigating Stable Chest Pain in Low to Intermediate Risk Women
Brief Title: Risk Evaluation and Stratification of Low Risk for Cardiovascular Disease in Women
Acronym: RESOLVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Elsie Nguyen (Other)
Responsible Party: Sponsor-Investigator, Elsie Nguyen, Associate Professor of Radiology, Women's College Hospital
Organization: Women's College Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-0069-B
Record Dates: First submitted 2019-01-15; First posted 2019-04-26 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Chest Pain
Keywords: angina
MeSH Terms: conditions — Chest Pain; Angina Pectoris

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CCTA first approach with Cardiac Link (Experimental): Patient will undergo Coronary Computed Tomography Angiography as the first test and have Cardiac Link pathway activated for expedited cardiology referral.
  Interventions: Diagnostic Test: Coronary Computed Tomography Angiography (CCTA); Other: Cardiac Link
- CCTA first approach without Cardiac Link (Experimental): Patient will undergo Coronary Computed Tomography Angiography as the first test, but Cardiac Link pathway will not be activated.
  Interventions: Diagnostic Test: Coronary Computed Tomography Angiography (CCTA)
- Usual Care with Cardiac Link (Active Comparator): Patient will undergo the usual diagnostic test ordered by their family physician as the first test, and have Cardiac Link pathway activated for expedited cardiology referral.
  Interventions: Diagnostic Test: Coronary Computed Tomography Angiography (CCTA); Other: Cardiac Link
- Usual Care without Cardiac Link (Active Comparator): Patient will undergo the usual diagnostic test ordered by their family physician as the first test, but Cardiac Link pathway will not be activated.
  Interventions: Diagnostic Test: Coronary Computed Tomography Angiography (CCTA)

INTERVENTIONS:
Diagnostic Test: Coronary Computed Tomography Angiography (CCTA) — Cardiac imaging test that is able to detect changes is cardiac vessels and the heart.
Other: Cardiac Link — Clinical patient flow pathway that will enable radiologist to activate expedited cardiology referral for patients who exhibit clinically significant changes during CCTA.
  Arms: CCTA first approach with Cardiac Link; Usual Care with Cardiac Link

SUMMARY:
This study will evaluate the ability of Coronary Computed Tomography Angiography (CCTA), used as a first-line diagnostic tool in women with stable chest pain and low risk for Coronary Artery Disease (CAD), to reduce the number of women requiring more than one diagnostic test to rule in or rule out CAD. Half of the participants will undergo CCTA as the first test to investigate stable chest pain, while the other half will undergo any test ordered by their family physician.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is the leading cause of death in women globally. Women are more likely to present with atypical chest pain that may be difficult to diagnose using traditional testing methods, resulting in over-investigation.

Coronary computed tomography angiography (CCTA) has high negative predictive value for exclusion of CAD in low to intermediate risk populations. We plan to investigate CCTA as a first line test to exclude coronary artery disease as a cause of stable chest pain and whether it is a cost effective strategy that reduces time to diagnosis, wait times to see cardiologists, emergency department visits, downstream and repeat testing and radiation exposure as compared to usual care with comparable patient safety and satisfaction level.

Another intervention being tested in this trial is the Cardiac Link pathway. This is a new clinical program at Women's College Hospital that aims to expedite cardiology referral for patients exhibiting clinically significant findings while undergoing CCTAs.

We hope that with use of CCTA as the first test, the number of women who require only one test (i.e. CCTA) to sort out whether or not CAD is responsible for their chest pain will increase, thereby decreasing over-investigation of low risk women.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age ≥ 40 years of age
* Stable chest pain or equivalent symptoms
* Planned non-urgent, non-invasive testing for diagnosis of chest pain or equivalent symptoms

Exclusion Criteria:

* Acute coronary syndrome, including acute myocardial infarction or unstable angina, known non-ischemic cardiomyopathy or other cardiac disease (e.g. mitral valve prolapse, etc.) which would require urgent cardiac evaluation
* Known CAD
* Prior cardiac evaluation for current episode of symptoms
* Previously investigated for CAD in the last 12 months
* Severe allergic reaction to iodinated contrast (mild reactions such as urticaria that can be controlled by premedication with Benadryl & Prednisone may be included in the study)
* Renal failure or dysfunction (estimated Glomerular Filtration Rate<30ml/min/m2 within the past 3 months)
* Pregnancy (status will be confirmed verbally. For premenopausal patients who are unsure, status will be confirmed by completing a pregnancy strip test).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2019-01-24 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Total Number of Tests | Through study completion, which may take up to 1 year
  The total number of tests a patient has to complete in order to diagnose the cause of their chest pain or equivalent symptoms

SECONDARY OUTCOMES:
Time to Diagnosis | From date of first presentation with chest pain to date of CAD diagnosis or exclusion, assessed up to 24 months
  Time interval from time of presentation to family physician for evaluation of chest pain to the last test performed to determine etiology of chest pain or CAD exclusion.
Wait Times to See a Cardiologist | From date of cardiology referral letter sent by family physician to date of cardiologist appointment with patient, assessed up to 24 months
  Time interval from when family physician referral letter was sent to the cardiologist's office to appointment time to see cardiologist
Hospital/ER visits | Through study completion, which may take up to 1 year
  Number of hospital/ER visits while waiting to see cardiologist
Number of Normal Invasive Diagnostic Angiograms | From date of randomization to date of CAD diagnosis or exclusion, assessed up to 24 months
  Number of invasive diagnostic angiograms done that reveal no coronary artery disease.
Total Cost of Investigations | Through study completion, which may take up to 1 year
  Total cost (in Canadian dollars) of all tests completed to reach a diagnosis for chest pain
Cumulative Radiation Dose Exposure (milliSieverts) | From date of randomization to date of CAD diagnosis or exclusion, assessed up to 24 months
  Total effective radiation dose from all testing modalities for each patient.

OTHER OUTCOMES:
Incidence of Procedure Related Adverse Events | From date of randomization to date of CAD diagnosis or exclusion, assessed up to 24 months
  Assessment of diagnostic procedure related adverse effects that may occur during the course of the trial.
Incidence of Cardiovascular Events | From date of randomization to date of CAD diagnosis or exclusion, assessed up to 24 months
  Assessment of cardiovascular events that may take place during the course of the study, while waiting for a diagnosis for the cause of chest pain

CONTACTS AND LOCATIONS:
Overall Officials: Elsie T Nguyen, MD, FRCPC, Principal Investigator — Women's College Hospital
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No